CLINICAL TRIAL: NCT04335162
Title: Cardiovascular Complications in Patients With COVID-19
Brief Title: Cardiovascular Complications and COVID-19 (CovCardioVasc-Study)
Acronym: CovCardioVasc
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20reamedcovid01
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: COVID; Acute Coronary Syndrome; Myocardial Infarction; Myocarditis; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocarditis; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with cardiovascular complications: Patients presenting with cardiomyopathies or venous thromboembolism
- Patients without cardiovascular complications: Patients without cardiomyopathies or venous thromboembolism
- Intensive Care Unit patients: Patients admitted in intensive care unit
- Hospital Ward patients: Patients admitted in hospital ward

SUMMARY:
Patients with COVID-19 in the Intensive Care Unit (ICU) or hospitalized with severe form have a poor prognosis (almost 30% rate of death). They present often a high cardiovascular risk profile (almost 30% of hypertension and 19% of diabetes). Troponin has been described to be elevated in a high proportion of patients (one fifth of all patients and 50% of non-survivors) suggesting the possibility of cardiomyopathies. High levels of DDimers (81% of non survivors) and fibrin degradation products are also associated with increased risk of mortality suggesting also the possibility of venous thromboembolism. Therefore, screening for cardiomyopathies and venous thromboembolism could represent an important challenge for patients with COVID-19 management.

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients with COVID-19 infection admitted to the ICU or hospitalized because of severe form (eg: hypoxia, orthopnea, pneumonitis, kidney insufficiency) will be included

Exclusion Criteria:

- Patients under 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intensive care unit, hospital ward
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Determine the incidence of cardiomyopathies and venous thromboembolism | 28 days
  Incidence of cardiomyopathies and/or venous thromboembolism at day 28

SECONDARY OUTCOMES:
Mortality | 28 days
  Incidence of mortality at day 28
Duration of mechanical ventilation | hospitalisation duration
  Number of day of using mechanical ventilation for each patients
Shock | hospitalisation duration
  Incidence of shock during hospitalisation
length of stay | hospitalisation duration
  Number of day at hospital
Mechanical ventilation | hospitalisation duration
  Setting up or not of mechanical ventilation
Renal replacement therapy | hospitalisation duration
  Administration or not of renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Denis DOYEN, Principal Investigator — CHU de NICE - Archet 1
Locations (8):
- France (8):
  - Centre Hospitalier de Cannes, Cannes
  - CHU de Dijon, Dijon
  - Centre Hospitalier de Draguignan, Draguignan
  - Centre Hospitalier de Grasse, Grasse
  - Clinique Ambroise-Paré, Neuilly
  - CHU de Nice, Nice
  - Hôpitaux Universitaires Paris Centre - Hôpital Cochin, Paris
  - CHU de REIMS, Reims

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established.

REFERENCES:
- [Derived] Jozwiak M, Dupuis C, Denormandie P, Aurenche Mateu D, Louchet J, Heme N, Mira JP, Doyen D, Dellamonica J. Right ventricular injury in critically ill patients with COVID-19: a descriptive study with standardized echocardiographic follow-up. Ann Intensive Care. 2024 Jan 23;14(1):14. doi: 10.1186/s13613-024-01248-8. PMID 38261092
- [Derived] Jozwiak M, Doyen D, Denormandie P, Goury A, Marey J, Pene F, Cariou A, Mira JP, Dellamonica J, Nguyen LS. Impact of sex differences on cardiac injury in critically ill patients with COVID-19. Respir Res. 2023 Nov 20;24(1):292. doi: 10.1186/s12931-023-02581-5. PMID 37986157
- [Derived] Ferrari E, Sartre B, Squara F, Contenti J, Occelli C, Lemoel F, Levraut J, Doyen D, Dellamonica J, Mondain V, Chirio D, Risso K, Cua E, Orban JC, Ichai C, Labbaoui M, Mossaz B, Moceri P, Appert-Flory A, Fischer F, Toulon P. High Prevalence of Acquired Thrombophilia Without Prognosis Value in Patients With Coronavirus Disease 2019. J Am Heart Assoc. 2020 Nov 3;9(21):e017773. doi: 10.1161/JAHA.120.017773. Epub 2020 Sep 25. PMID 32972320